CLINICAL TRIAL: NCT05145933
Title: Head Start REACH: Strengthening Outreach, Recruitment and Engagement Approaches With Families
Acronym: HSREACH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Boston Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 51075
Record Dates: First submitted 2021-10-29; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-09

CONDITIONS: Early Intervention, Educational (Head Start and Early Head Start Access and Participation)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mathematica, funded by the Administration for Children and Families (ACF) Office of Planning, Research, and Evaluation (OPRE) in the U.S. Department of Health and Human Services (HHS) will collect descriptive information for the Head Start REACH: Strengthening Outreach, Recruitment and Engagement Approaches with Families (Head Start REACH) study. The investigators will conduct qualitative case studies in six sites. The goal of these case studies in the Head Start REACH study is to provide an in-depth understanding of (1) the approaches that are likely to be successful for the recruitment, selection, enrollment, and retention (RSER) of families who are experiencing adversities; (2) the factors that affect the implementation of these approaches and; (3) the experiences of such families, both enrolled and non-enrolled in Head Start.

Data collection will occur in spring 2022. The investigators will conduct qualitative, semi-structured interviews with staff across the six sites who are involved in RSER efforts and provide services to families experiencing adversities, including those in Head Start programs and in the community organizations with which the programs partner. The investigators will also conduct focus groups with families who are being served by Head Start programs and/or the community partner organizations.

DETAILED DESCRIPTION:
This study aims to advance understanding of the approaches that programs use for the recruitment, selection, enrollment, and retention (RSER) of families who are experiencing adversities; the implementation of those approaches; and the experience of Head Start-eligible families (both enrolled and not enrolled in Head Start). Adversities is a broad term that refers to a wide range of circumstances or events that pose a threat to a child or caregiver's physical or psychological well-being. The adversities that families experience are often intertwined with poverty, may co-occur, and are affected by systematic factors, such as structural racism. Common examples include (but are not limited to) families experiencing homelessness; involvement in child welfare, including foster care; and affected by substance use, mental health issues, and domestic violence. Data from these case studies will inform the development of the study's conceptual framework, identify knowledge gaps, and inform the design of a future large-scale descriptive study. Ultimately, this information collection will support ACF in better understanding how Head Start programs recruit, select, enroll, and retain families and inform Head Start's efforts to achieve its mission of advancing equitable outcomes for children and families. In addition, these case studies may identify promising approaches for engaging underserved populations and help Head Start utilize more effective case management and coordination strategies.

The information collected is meant to contribute to the body of knowledge on ACF programs. It is not intended to be used as the principal basis for a decision by a federal decision-maker and is not expected to meet the threshold of influential or highly influential scientific information.

The investigators propose the following data collection activities, to be carried out in spring 2022:

1. A semi-structured program director interview: To obtain information about the Head Start program's eligibility, recruitment, selection, enrollment, and attendance (ERSEA) policies; RSER approaches and how they are tailored for families facing adversities; staff training and support related to RSER and adversities; RSER approaches used with underserved families; and partnerships that support the program's RSER efforts.
2. A semi-structured Head Start ERSEA staff interview: To obtain information about the Head Start program's ERSEA policies; RSER approaches and how they are tailored for families facing adversities; staff training and support related to RSER and adversities; RSER approaches used with underserved families; and partnerships that support the program's RSER efforts.
3. A semi-structured community partner staff interview: To collect information about the community organization's experience working with the Head Start program and their referral processes; the organization's understanding of Head Start eligibility criteria; the organization's procedures for disseminating information about early education and child care options to families; and the organization's view of the Head Start program's role in meeting families' needs.
4. A focus group with families enrolled in Head Start: To collect information on the families' experience with the Head Start program; the recruitment and post-enrollment experience in the Head Start program; and the likelihood of the family's continuing its involvement in the Head Start program.
5. A focus group with Head Start-eligible families not enrolled in Head Start: To obtain information on the families' experience with the community partner organization; knowledge of Head Start program and alternate early education and child care options; barriers to enrollment in the Head Start program; and the reasons families choose alternative child care.

ELIGIBILITY:
Inclusion Criteria:

* Program director at Head Start program
* ERSEA staff members at Head Start program
* Staff at community partner organizations
* Families enrolled in program at Head Start program
* Families not enrolled in Head Start program but being served by the community partner organization

Exclusion Criteria:

* Does not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Head Start program directors; Head Start staff involved in implementing eligibility, recruitment, selection, enrollment, and attendance (ERSEA) activities; staff in community organizations with which the Head Start program partners to serve families experiencing adversities; families who are enrolled in Head Start programs; and families who are eligible for but not enrolled in Head Start programs.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2022-01-03 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Program Staff Interview Protocol on Promising RSER Approaches: Program Director | 1 month
  Study developed qualitative protocol will collect data on Head Start program approaches used for the recruitment, selection, enrollment, and retention (RSER) of families facing adversities and report on the most promising RSER approaches.
Program Staff Interview Protocol on Promising RSER Approaches: ERSEA Staff | 1 month
  Study developed qualitative protocol will collect data on Head Start program approaches used for the RSER of families facing adversities and report on the most promising RSER approaches.
Focus Group Guide for Head Start Enrolled Families on Head Start Recruitment and Post-enrollment Experiences | 1 month
  Study developed qualitative protocol will collect data on the recruitment and post-enrollment experience of families experiencing adversities who are enrolled in Head Start programs and report on the factors that facilitate successful enrollment and retention of these families.
Community Partner Staff Interview Protocol on Factors that Support RSER | 1 month
  Study developed qualitative protocol will collect data and report on the factors that support the Head Start program's RSER of families experiencing adversities
Focus Group Guide for Families Not Enrolled in Head Start on Barriers to Head Start Participation | 1 month
  Study developed qualitative protocol will collect data on the experience of families experiencing adversities who are not enrolled in Head Start programs and report on the factors that prevent their participation.

CONTACTS AND LOCATIONS:
Locations (1):
- Mathematica, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Information about program-level respondents and respondents from community partner organizations will be kept private to the extent permitted by law; information about parents who participate in the focus groups will be kept private to the extent permitted by law. Any data shared for the project will be shared in summary form.